CLINICAL TRIAL: NCT00890487
Title: Effects of Hyaluronic Acid Oral Supplementation on the Vaginal Epithelium: a Prospective, Randomized, Double-Blind, Placebo Controlled Study
Brief Title: Hyaluronic Acid and Vaginal Distress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Messina (Other)
Responsible Party: G.Marino University Policlinic of Messina, Menopause centre of
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 30031978
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Vaginal Disease
MeSH Terms: conditions — Vaginal Diseases | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- hyaluroni acid pill (Other)
  Interventions: Other: hyaluronic acid pill

INTERVENTIONS:
Other: hyaluronic acid pill — pill, 220 mg, once a day, three months

SUMMARY:
The purpose of this trial is to study the effects of the oral supplementation hyaluronic acid in menopause women with vaginal distress for treatment vaginal distress.

ELIGIBILITY:
Inclusion Criteria:

* menopause
* vaginal distress
* no other therapy

Exclusion Criteria:

* vaginal infection
* Sjogren Syndrome

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-09 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
effects of the oral somministration hyaluronic acid in menopause women with vaginal distress | three months

CONTACTS AND LOCATIONS:
Overall Officials: Tindara TL La Galia, PhD student, Principal Investigator — Centre Menopause
Locations (1):
- Menopause centre of the G. Martino University Policlinic, Messina, Sicily, Italy